CLINICAL TRIAL: NCT00684762
Title: A Comparative Bioavailability Study of Cilostazol Tablets, 100mg Under Fasting Conditions
Brief Title: Fasted Bioavailability Study of Cilostazol Tablets, 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Kristin Arnold, Vice President R&D, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11788
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2009-12-22 (Estimated); Status verified 2009-11

CONDITIONS: Therapeutic Equivalency
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol (Experimental): A single dose of cilostazol (1 x 100 mg tablet) administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Cilostazol 100 mg Tablets
- Pletal® (cilostazol) (Experimental): A single dose of cilostazol (Pletal® 1 x 100 mg tablet) administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Cilostazol (Pletal®) 100 mg Tablets

INTERVENTIONS:
Drug: Cilostazol 100 mg Tablets — Cilostazol (1 x 100 mg tablet) administered after an overnight fast of at least 10 hours
  Arms: Cilostazol
Drug: Cilostazol (Pletal®) 100 mg Tablets — Cilostazol (Pletal® 1 x 100mg tablet) administered after an overnight fast of at least 10 hours.
  Other Names: Pletal®
  Arms: Pletal® (cilostazol)

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability of a test formulation of cilostazol tablets to an equivalent dose of Pletal® (cilostazol) tablets after a single oral dose administered under fasting conditions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability of a test formulation of cilostazol tablets to an equivalent dose of Pletal® (cilostazol) tablets after a single oral dose administered under fasting conditions. Thirty-two non-smoking, non-obese, healthy male and female volunteers between the ages of 18 and 55 will be randomly assigned in a crossover fashion to receive each of two cilostazol dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will receive either a single oral dose of the test formulation, cilostazol (1 x 100 mg tablet), or a single oral dose of the reference formulation, Pletal® (1 x 100 mg tablet). After a 7 day washout period on the morning of Day 8, following an overnight fast of at least 10 hours, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of cilostazol. Blood sampling will then continue on a non-confined basis at 36 and 48 hours post-dose. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. Blood pressure and pulse will be measured before dosing and at 3 and 24 hours post-dose. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-55 years of age
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* No more than 15% plus or minus from ideal weight for subject's height and elbow breadth as defined by the Metropolitan Life Insurance Company Statistical Bulletin. Extrapolations, if required, to be conducted according to BASi Standard Operating Procedures
* Medically healthy on the basis of medical history and physical examination within 30 days prior to the start of the study
* Test results from blood chemistry, hematology, and urinalysis performed within 30days prior to the start of the study within clinically acceptable limits
* At screening, subjects must have blood pressure and pulse rate within the following ranges: Systolic blood pressure 90-140mmHg; Diastolic blood pressure 50-90mmHg; Pulse 45-100 bpm
* An acceptable electrocardiogram (EKG): sinus rhythm with no evidence of AV block or ischemic changes

Exclusion Criteria:

* Prescription drug use (excluding hormonal contraceptives) within 14 days prior to drug administration, each period
* Aspirin ingestion within 7 days prior to drug administration, each period
* Use of any over-the-counter preparations, herbal remedies, and/or nutritional supplements within 7 days prior to drug administration, each period
* Consumption of grapefruit juice or grapefruit-containing products within 72 hours prior to drug administration , each period
* Consumption of alcohol within 24 hours prior to drug administration, each period
* Consumption of caffeine within 10 hours prior to drug administration, each period
* Female subjects must not be pregnant or nursing; and must be surgically sterile; one year post-menopausal; or on hormonal contraceptive agent(s), a diaphragm or condom with spermicidal foam or jelly, or IUD for at least three months prior to drug administration and agree to use the same method of contraception for at least 1 month after the last drug administration
* Subjects with a history or presence of significant organ system (cardiovascular, neurological, hepatic, hematopoietic, renal, pulmonary, endocrine, or gastrointestinal) disorders, or ongoing infectious diseases
* History of hypersensitivity or adverse reactions to cilostazol (Pletal®), or other related drugs
* Recent (12 month) history or evidence of alcoholism or drug abuse
* Positive results to Human Immunodeficiency Virus (HIV) or Hepatitis B surface Antigen (HBsAg) tests

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilip K Guha-Ray, M.D., Principal Investigator — BASi Baltimore Clinical Research Unit

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cilostazol 100 mg Tablets Then Pletal® 100 mg Tablets: On the morning of Day 1 subjects received one tablet of the test formulation, Cilostazol 100 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received one tablet of the reference formulation, Pletal® 100 mg, after an overnight fast of at least 10 hours.
- Pletal® 100 mg Tablets Then Cilostazol 100 mg Tablets: On the morning of Day 1 subjects received one tablet of the reference formulation, Pletal® 100 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received one tablet of the test formulation, Cilostazol 100 mg, after an overnight fast of at least 10 hours.
Period: First Intervention
Arm/Group | Cilostazol 100 mg Tablets Then Pletal® 100 mg Tablets | Pletal® 100 mg Tablets Then Cilostazol 100 mg Tablets
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Cilostazol 100 mg Tablets Then Pletal® 100 mg Tablets | Pletal® 100 mg Tablets Then Cilostazol 100 mg Tablets
Started | 16 | 16
Completed | 14 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Second Intervention
Arm/Group | Cilostazol 100 mg Tablets Then Pletal® 100 mg Tablets | Pletal® 100 mg Tablets Then Cilostazol 100 mg Tablets
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cilostazol 100 mg Tablets and Pletal® 100 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either Cilostazol 100 mg or Pletal® 100 mg following an overnight fast of at least 10 hours.
Arm/Group | Cilostazol 100 mg Tablets and Pletal® 100 mg Tablets
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.09 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that cilostazol (test and reference product) reaches in the plasma.
Time Frame: serial pharmacokinetic concentrations were drawn pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 16, 24, 36 and 48 hours post-dose.
Population: Plasma concentration data for 28 of the 32 enrolled participants were used in the statistical analysis. Four subjects did not complete the study and none of their collected data was used.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cilostazol 100 mg Tablets: On the morning of Day 1 subjects received one tablet of either the test formulation, cilostazol 100mg, or the reference formulation, Pletal® 100 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received the alternate regimen following an overnight fast of at least 10 hours.
- Pletal® 100 mg Tablets: On the morning of Day 1 subjects received one tablet of the reference formulation, Pletal® 100 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received one tablet of the test formulation, Cilostazol 100 mg, after an overnight fast of at least 10 hours.
Arm/Group | Cilostazol 100 mg Tablets | Pletal® 100 mg Tablets
Number analyzed (Participants) | 28 | 28
ng/mL | 484.895 (205.181) | 472.689 (140.843)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable cilostazol (test and reference) concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Cilostazol 100 mg Tablets | Pletal® 100 mg Tablets
Number analyzed (Participants) | 28 | 28
ng-hr/mL | 6,518.90 (1,600.14) | 6,711.57 (1,895.25)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable cilostazol (reference and test) plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Plasma concentration data for 26 of the 32 enrolled participants were used in the statistical analysis. Four subjects did not complete the study and none of their collected data was used. Additionally, two subjects had data values that were not used in this analysis.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Cilostazol 100 mg Tablets | Pletal® 100 mg Tablets
Number analyzed (Participants) | 26 | 26
ng-hr/mL | 7,224.99 (1,786.61) | 7,650.45 (2,294.39)

ADVERSE EVENTS:
Description: 32 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving both interventions. 30 subjects were administered cilostazol 100 mg tablets and 30 subjects were administered Pletal® 100 mg tablets.
Groups:
- Cilostazol 100 mg Tablets; Pletal® 100 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either cilostazol 100 mg or Pletal® 100 mg following an overnight fast of at least 10 hours.
Arm/Group | Cilostazol 100 mg Tablets | Pletal® 100 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/30 | 12/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol 100 mg Tablets (N=30) | Pletal® 100 mg Tablets (N=30)
Headache (Nervous system disorders) | 6 (6) | 6 (6)
Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Pain and burning post venipuncture
Eosinophilia (Investigations) | 0 (0) | 1 (1) — Increased levels of eosinophils in blood
Lymphadeno (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — swollen glands left lateral neck with jaw angle; pain on swallowing
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Elevated level of glucose in blood
LDH increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Elevated LDH level in blood
SGOT increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Elevated SGOT level in blood
Paresthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Numbness and tingling in left hand and forearm post phlebotomy
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Nasal congestion
Urine abnormal (Renal and urinary disorders) | 0 (0) | 3 (3) — Elevated levels of leukocyte esterase U/A; Elevated levels of WBC/HPF in U/A as well as leukocyte esterase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days